Statistical Analysis Plan

29 November 2016, Version 1.0



# STATISTICAL ANALYSIS PLAN

**Title** An Open-Label, Phase 2 Study to Assess the Safety,

> Pharmacodynamics, and Efficacy of KRN23 in Children from 1 to 4 Years Old with X-linked Hypophosphatemia

(XLH)

**Protocol:** UX023-CL205

**Investigational Product:** KRN23 (Recombinant human IgG1 monoclonal antibody

to fibroblast growth factor 23 [FGF23])

Phase: 2

Ultragenyx Pharmaceutical Inc. **Sponsor:** 

60 Leveroni Court

Novato, CA, USA 94949

PhD **Author:** 

Manager, Biostatistics, Biometrics

29 November 2016 Date:

**Version Number:** 1.0



# **TABLE OF CONTENTS**

| 1 | INT | RODUCTION7 |
|---|-----|------------------------------------|
| 2 | STU | DY OBJECTIVE(S)8 |
| | 2.1 | Primary Objective |
| | 2.2 | Other Objective |
| 3 | STU | DY DESIGN9 |
| | 3.1 | Study Population9 |
| | 3.2 | Dosage and Administration9 |
| | 3.3 | Blinding and Randomization Methods |
| | 3.4 | Stratification Factors |
| | 3.5 | Sample Size Considerations |
| | 3.6 | Planned Analyses |
| | 3.7 | Data Monitoring Committee |
| 4 | STU | DY ENDPOINTS, COVARIATES11 |
| | 4.1 | Primary Efficacy Endpoints |
| | 4.2 | Secondary Efficacy Endpoints |
| | 4.3 | Other Efficacy Endpoints |
| | 4.4 | Safety Endpoints |
| | 4.5 | Drug Concentration Measure |
| | 4.6 | Covariate(s)12 |
| 5 | DEF | INITIONS |
| | 5.1 | Baseline |
| | 5.2 | Study Day13 |
| | 5.3 | Age13 |
| | 5.4 | RGI-C13 |
| | 5.5 | RSS |
| | 5.6 | Growth |



| | | 5.6.1 | Standing height/recumbent length Z-score and Percentile | 15 |
|---|---|---|---|---|
| | | 5.6.2 | Weight Z-score and Percentile | 16 |
| | 5.7 | Blood I | Pressure Percentile | 16 |
| | 5.8 | Heart R | ate Percentile | 16 |
| | 5.9 | Events | to Monitor | 16 |
| | 5.10 | Dose L | imiting Toxicity | 17 |
| | 5.11 | Duratio | n of SOC | 17 |
| 6 | ANA | ALYSIS | POPULATIONS | 18 |
| | 6.1 | Efficac | y Analysis Set | 18 |
| | 6.2 | Safety A | Analysis Set | 18 |
| | 6.3 | Pharma | cokinetic (PK) and Pharmacodynamic (PD) Analysis Set | 18 |
| 7 | DAT | CA SCRI | EENING AND ACCEPTANCE | 19 |
| | 7.1 | Genera | Principles | 19 |
| | 7.2 | Handlir | ng of Missing and Incomplete Data | 19 |
| | | 7.2.1 | Missing Date Information for Adverse Events and Concomitant<br>Medications | 19 |
| | | 7.2.2 | Missing Causal Relationship to Investigational Product for Adverse Events | 20 |
| | 7.3 | Unsche | duled and Early Termination Visits | 20 |
| | 7.4 | Softwar | ·e | 20 |
| 8 | STA | TISTIC | AL METHODS OF ANALYSES | 21 |
| | 8.1 | Genera | Principles | 21 |
| | 8.2 | Subject | Accountability | 21 |
| | 8.3 | Protoco | l Deviations | 21 |
| | 8.4 | Investig | gational Product Administration | 21 |
| | 8.5 | Demog | raphic and Baseline Characteristics | 21 |
| | 8.6 | Prior ar | nd Concomitant Medication | 22 |
| | 8.7 | Medica | l History / XLH Medical and Family History | 22 |



| 8.8 | Efficac | y Analysis | 22 |
|---|---|---|---|
| | 8.8.1 | Generalized Estimating Equations Model | 22 |
| | 8.8.2 | Primary Efficacy Endpoint | 23 |
| | 8.8.3 | Secondary Efficacy Endpoints | 23 |
| | | 8.8.3.1 RGI-C | 23 |
| | | 8.8.3.2 RSS | 23 |
| | | 8.8.3.3 Growth | 24 |
| | 8.8.4 | Other Pharmacodynamics Parameters | 24 |
| 8.9 | Pharma | acokinetics | 24 |
| 8.10 | Safety | Analysis | 24 |
| | 8.10.1 | Adverse Events | 24 |
| | 8.10.2 | Safety Lab Parameters | 25 |
| | 8.10.3 | Physical Examination | 25 |
| | 8.10.4 | Vital Signs | 25 |
| | 8.10.5 | Renal Ultrasound | 25 |
| | 8.10.6 | Electrocardiogram | 26 |
| 9 REF | ERENC | ES | 27 |
| 10 APP | ENDIC | ES | 28 |
| List of T | Γables | | |
| Table 8. | 10.6.1: | Criteria for ECG Results | 26 |
| Table 10 | ).1: | Schedule of Events – Screening, Baseline, and Treatment Period Weeks 1-30 | 31 |
| Table 10 | 0.2: | Schedule of Events – Treatment Period Weeks 32 – 64 | 33 |



# **List of Appendices**

| Appendix 1: | Efficacy Endpoint Summary Table | 28 |
|---|---|---|
| Appendix 2: | Clinical Laboratory Assessments for Safety | 29 |
| Appendix 3: | Schedule of Events | 31 |
| Appendix 4: | RSS Data Collection Form | 36 |
| Appendix 5: | RGI-C Data Collection Form | 38 |
| Appendix 6: | Blood Pressure Percentiles by Gender, Age and Height (NHLBI 2005) | 42 |
| Appendix 7: | Heart Rate Percentiles by Gender and Age | <b>4</b> 4 |
| Appendix 8: | Events to Monitor | 45 |

Statistical Analysis Plan 29 November 2016, Version 1.0



## **ABBREVIATIONS**

1,25(OH)<sub>2</sub>D 1,25-dihydroxyvitamin D

AE Adverse Event

ALP Alkaline Phosphatase

BP Blood Pressure

CRF Case Report Form

CDC/NCHS Centers for Disease Control/National Center for Health Statistics

EDC Electronic Data Capture

eGFR Estimated Glomerular Filtration Rate

iPTH Intact Parathyroid Hormone

IP Investigational Product
ISR Injection Site Reaction

HAHA Human Anti-Human Antibody

HR Heart Rate

HLT High-Level Term

MedDRA Medical Dictionary for Regulatory Activities

PD Pharmacodynamic(s)
PK Pharmacokinetic(s)
RR Respiratory Rate

RSS Rickets Severity Score SAE Serious Adverse Event

SAP Statistical Analysis Plan

SOC Standard of Care

TEAE Treatment-Emergent Adverse Event

TESAE Treatment-Emergent Serious Adverse Event

XLH X-linked Hypophosphatemia




# 1 INTRODUCTION

The purpose of this Statistical Analysis Plan (SAP) is to provide details of the statistical analyses that have been outlined within the UX023-CL205 Protocol Amendment 1 dated 28 March 2016. The SAP for Week 4 analysis was pre-specified in a separate document (UX023-CL205 Statistical Analysis Plan Week 4 Analysis) before the analysis took place.




# 2 STUDY OBJECTIVE(S)

## 2.1 Primary Objective

The primary objectives of the study are to:

- Establish the safety profile of KRN23 for the treatment of XLH in children between 1 and 4 years old
- Determine the PD effects of KRN23 treatment on serum phosphorus and other PD markers that reflect the status of phosphate homeostasis in children between 1 and 4 years old with XLH

# 2.2 Other Objective

Additional study objectives are to assess the following in children between 1 and 4 years old with XLH:

- Effects of KRN23 on rickets
- Effects of KRN23 on growth and lower extremity deformity
- Pre-dose KRN23 drug concentration levels




## 3 STUDY DESIGN

As background for the statistical methods presented below, this section provides an overview of the study design. This overview is a summary only. The protocol is the definitive reference for all matters discussed in what follows.

## 3.1 Study Population

UX023-CL205 is a multicenter, open-label, Phase 2 study in children from 1 to 4 years old with XLH who are naïve to therapy or have previously received standard therapy with oral phosphate and active vitamin D to assess the safety, PD, and efficacy of KRN23 administered via subcutaneous injections Q2W for a total of 64 weeks.

## 3.2 Dosage and Administration

The length of this study will be 64 weeks. All subjects will receive KRN23 at a starting dose of 0.8 mg/kg every two weeks (Q2W). The dose may be increased to 1.2 mg/kg at any time if a subject meets the following dose adjustment criteria: 1) two consecutive serum phosphorus measurements are below the normal range; 2) serum phosphorus has increased by < 0.5 mg/dL from baseline; and 3) the subject has not missed a dose of study drug that would account for the decrease in serum phosphorus.

At any time during the study, if serum phosphorus increases above the upper limit of normal for age, the subsequent dose(s) will be withheld and the site will contact the medical monitor before dosing resumes. Once other causes of increased serum phosphorus are excluded, KRN23 treatment will resume at half the total dose of the last dose received. Serum phosphorus will be followed through unscheduled serum phosphorus assessments. A subject will resume dosing at the previous full total dose level if they meet the same dose-adjustment criteria listed above.

Serum phosphorus assessments will be conducted at the clinic at the ends of Weeks 1, 4, 8, 12, 15, 20, 32, 40, 48, 56 and 64. Growth (recumbent length/standing height) assessment will be conducted at the ends of Week 12, 24, 40 and 64. Bilateral AP knee X-rays, bilateral PA hand/wrist X-rays and standing long leg X-rays will be conducted at Week 40 and 64. The schedule of assessments is shown in Appendix 3.

## 3.3 Blinding and Randomization Methods

The UX023-CL205 is an open-label Phase 2 study; all subjects will receive same starting dose Q2W. Blinding or randomization methods are not applicable for this study.

#### 3.4 Stratification Factors

Stratification factors are not applicable for this study.




# 3.5 Sample Size Considerations

The study will enroll approximately 10 pediatric subjects between 1 and 4 years old, inclusive, with clinical findings consistent with XLH including hypophosphatemia and radiographic evidence of rickets (at least 5 subjects will have a rickets severity score (RSS) at the knee of  $\geq$ 1.5 points at Screening), and a confirmed *PHEX* mutation or variant of uncertain significance. To maintain a level of gender balance, no more than 7 subjects of either gender will be enrolled.

# 3.6 Planned Analyses

The primary analysis is planned at Week 40. Additional efficacy and safety analyses will be conducted at Week 64. A Week 24 analysis has been planned as an administrative analysis to support regulatory interaction. The analysis will include safety, Pharmacokinetics (PK), Pharmacodynamics (PD), and growth assessments; rickets assessment from radiographs will not be included as the radiographs are not scheduled until Week 40. Additional administrative analyses may be done at the sponsor's discretion to support regulatory submission or product planning.

## 3.7 Data Monitoring Committee

An independent DMC that includes members with expertise in metabolic bone disease, cardiology, nephrology, and the conduct of clinical trials in children will act in an advisory capacity to monitor subject safety on a routine basis throughout the trial. The DMC will meet approximately twice a year. The roles and responsibilities of the DMC will be defined in the DMC Charter.




#### 4 STUDY ENDPOINTS, COVARIATES

All data are collected according to the schedule of assessments (Appendix 3).

## 4.1 Primary Efficacy Endpoints

The primary efficacy endpoint is the change from baseline in serum phosphorus.

# 4.2 Secondary Efficacy Endpoints

The secondary efficacy endpoints include

- Change in rickets at Week 40 as assessed by the Radiograph Global Impression of Change (RGI-C) global score
- Change in rickets at Week 64 as assessed by RGI-C global score
- Change from baseline in Rickets Severity Score (RSS) total score at Weeks 40 and 64
- Change in lower extremity skeletal abnormalities, including genu varum and genu valgus, as determined by the RGI-C long leg score at Weeks 40 and 64
- Change in recumbent length/standing height from baseline to post-treatment study time points in cm, height-for-age z-scores, and percentiles. Historical growth records may be used to evaluate change in growth velocity
- Change and percent change from baseline over time in serum alkaline phosphatase (ALP)

# 4.3 Other Efficacy Endpoints

Other efficacy endpoints include

- Change from baseline over time in serum 1,25(OH)<sub>2</sub>D and urinary phosphorus
- Change in rickets at Week 40 and 64 as assessed by RGI-C wrist score and knee score
- Change from baseline in RSS wrist score and knee scores at Week 40 and 64

#### 4.4 Safety Endpoints

General Safety Variables will include the following:

- Treatment Emergent Adverse Events (TEAEs)
- Treatment Related TEAEs
- Treatment Emergent Serious Adverse Events (TESAEs)
- Events to monitor:
  - Injection site reaction (High-Level Term)
  - Immunogenicity




- Hyperphosphatemia
- Ectopic mineralization
- Restless leg syndrome
- Grade 3/4 TEAEs
- TEAEs leading to discontinuation from the study
- TEAEs leading to discontinuation from the study drug treatment
- TEAEs leading to death
- Vital signs and weight
- Physical examinations
- Estimated Glomerular Filtration Rate (eGFR)
- Chemistry, hematology, and urinalysis, including additional KRN23/XLH biochemical parameters of interest (serum calcium, intact parathyroid hormone[iPTH], 25-hydroxyvitamin D [25(OH)D], amylase, lipase, and creatinine; and urinary calcium and creatinine)
- FGF23
- Anti-KRN23 antibody (HAHA) testing and Dose-Limiting Toxicities (DLT)
- Concomitant medications

Ectopic Mineralization Safety Assessments include:

- Renal ultrasound
- Electrocardiogram (ECG)

## 4.5 Drug Concentration Measure

To assess KRN23 concentration and possible accumulation, serum pre-dose levels will be evaluated as a PK parameter in this study.

#### 4.6 Covariate(s)

Baseline measures will be used as covariates. For example, baseline RSS score will be used in the modeling for change in baseline in RSS score and for RGI-C score. Age and gender may also be used as covariates in growth endpoint models.




#### 5 DEFINITIONS

#### 5.1 Baseline

Baseline is defined as the last assessments prior to or on the date of initiation of the first dose of investigational product.

## 5.2 Study Day

Study day is calculated as:

(visit date – date of the first dose of investigational product + 1) if the visit data is on or after the first dose of investigational product; or (visit date – date of the first dose of investigational product) if the visit data is prior the first dose of investigational product.

## **5.3** Age

Unless specified, the age will be derived based on the informed consent date: Age =  $(Informed\ Consent\ Date\ -\ Birth\ Date\ +1)/365.25$ . The age will be rounded down to the nearest x.x years and keep one decimal place.

#### **5.4 RGI-C**

Changes in the severity of rickets and bowing will be assessed centrally by three independent pediatric radiologists contracted by a central imaging facility using a disease specific qualitative Radiographic Global Impression of Change (RGI-C) scoring system.

The RGI-C is a seven point ordinal scale with possible values:

- +3 = very much better (complete or near complete healing of rickets),
- +2 = much better (substantial healing of rickets),
- +1 = minimally better (i.e., minimal healing of rickets),
  - 0 = unchanged,
- -1 = minimally worse (minimal worsening of rickets),
- -2 = much worse (moderate worsening of rickets),
- -3 = very much worse (severe worsening of rickets),

Raters will be presented with side-by-side images taken from subjects during the UX023-CL205 study with the Baseline image on the left (Image A) and Post-Treatment image (Week 40 and Week 64) on the right (Image B). Raters will be asked to evaluate change in Image B for the abnormalities they consider to be present in the Baseline Image A. This exercise will be performed for the distal radius and ulna from the bilateral wrist X-rays, and the distal femur and proximal tibia and fibula from the bilateral knee X-rays at Week 40 and Week 64. At Week 64, Image A (presented on the left) will remain the Baseline image and Image B (presented on the right) will be the post-treatment image from Week 64.




In addition to bilateral wrists and knees, the Week 40 and Week 64 RGI-C analysis will include a rating of the full femur, tibia and fibula from the bilateral standing long leg film with the Baseline standing long leg image on the left (Image A) and the Week 40 (or Week 64) standing long leg image on the right (Image B). The RGI-C is scored using a pre-defined methodology (Biomedical Systems Independent Review Manual July 2015). See data collection form in Appendix 5.

Prior to rating, the three raters will be trained to gain consensus on the terminology used to describe XLH-related radiographic abnormalities and to establish inter-rater reliability. Following the training, each rater will independently complete a quiz involving the rating of practice images to ensure the success of the training and the reliability of scores among the raters. For the Week 40 and Week 64 analysis, each of the three raters will perform the rating exercise at a work station at the central imaging facility. Only one rater can be present at the facility at any given time to prevent group rating or sharing of scores. Each rater will be presented with side-by-side images of the wrist and knee with Baseline on the left (Image A) and Post-Treatment on the right (Image B). Raters will be asked to evaluate the presence of various abnormalities in the wrist and knee in Image A and change in those abnormalities in Image B. At the Week 40 and Week 64 analysis, each rater will evaluate changes in rickets severity from Baseline to Week 40 in the wrists and knees by assigning a regional score for the wrist, a regional score for the knee, as well as an overall impression score (RGI-C global score). The RGI-C scores for the three raters will be averaged and the mean scores for the wrist, knee and overall impression will be reported. The raters will also evaluate images from long leg radiographs. The RGI-C scores from the three raters will be averaged to generate a RGI-C lower limb deformity score. RGI-C scores will be entered into an EDC system at the time of the scoring and cannot be retrieved or changed by the rater after submission. RGI-C scores will be transferred electronically from the imaging facility to Ultragenyx after the image rating exercise is complete.

RGI-C response is defined as an averaged RGI-C global score of at least +2.0 (i.e. substantial healing of rickets).

#### 5.5 RSS

The severity of rickets will be measured using a scale developed by Thomas Thacher, MD for the assessment of nutritional rickets (Thacher et al. 2000). This scale will be referred to as the RSS. The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points, with a total possible score of 4 points for the wrists and 6 points for the knees. Higher scores indicate greater rickets severity. The RSS is scored using a pre-defined methodology (Biomedical Systems Independent Review Manual September 2014). Each radiograph is scored individually by Dr. Thacher who will serve as the single central independent rater for all UX023-CL205 X-rays taken at Baseline, Week 40 and Week 64. For the X-rays taken during the




UX023-CL205 study, Dr. Thacher will be blinded to the study visit at which the X-ray was taken, adherence to the study protocol and duration of treatment. Each rating performed by Dr. Thacher is entered into an EDC system at the time of the rating and transferred electronically to a central imaging facility. The scores cannot be retrieved from the system by Dr. Thacher after submission. See RSS data collection form in Appendix 4.

#### 5.6 Growth

## 5.6.1 Standing height/recumbent length Z-score and Percentile

Recumbent length will be measured in subjects < 2 years old or those unable or unwilling to stand for the measurement. Standing height/recumbent length measurements prior to treatment will be abstracted from medical records where available.

Growth as measured by standing height or recumbent length will be evaluated on a percentile basis using the Centers for Disease Control/National Center for Health Statistics (CDC/NCHS) Clinical Growth Charts (Kuczmarski et al. 2000). Data used to produce the United States Growth Charts smoothed percentile curves will be downloaded from the official CDC/NCHS web site: http://www.cdc.gov/growthcharts/percentile\_data\_files.htm

The data files from the CDC/NCHS that are used for this analysis are summarized below. These files represent the different growth curves for children. LMS refers to the parameters in the CDC Growth Charts Percentile Data Files used to construct the growth curves; these are: the power in the Box-Cox transformation (L); the median (M); and the generalized coefficient of variation (S).

The data files used are:

- Length-for-age charts, birth to 36 months, LMS parameters and selected smoothed recumbent length percentiles in centimeters, by sex and age (LENAGEINF).
- Stature-for-age charts, 2 to 20 years, LMS parameters and selected smoothed stature percentiles in centimeters, by gender and age (STATAGE).

Calculation of Z-scores for length/stature values above and below the median will be performed. Using the CDC/NCHS Clinical Growth Charts, the height-for-age Z score will be calculated using the following equation:

$$Z = \{(X/M)^{L} - 1\} / (L \times S),$$

where X is the physical measurement (stature in cm) and the LMS parameters are obtained from the appropriate CDC/NCHS Clinical Growth Chart corresponding to the age in months of the child. The percentile corresponding to the Z score is then the corresponding percentile from the standard normal distribution.




# 5.6.2 Weight Z-score and Percentile

Weight will be evaluated by z score and percentile using the same method as Section 5.7.1 based on Centers for Disease Control/National Center for Health Statistics (CDC/NCHS) Clinical Growth Charts (Kuczmarski et al. 2000). The data files used for weight Z-score and percentile are:

- Weight-for-age charts, birth to 36 months, LMS parameters and selected smoothed weight percentiles in kilograms, by sex and age (WTAGEINF).
- Weight-for-age charts, 2 to 20 years, LMS parameters and selected smoothed weight percentiles in kilograms, by sex and age (WTAGE).

## **5.7** Blood Pressure Percentile

The blood pressure percentile will be derived based on the Fourth Report on the Diagnosis, Evaluation and Treatment of High Blood Pressure in Children and Adolescents (NHLBI 2005). See Appendix 6 for details in deriving blood pressure percentile adjusting for age, gender and height.

## 5.8 Heart Rate Percentile

The heart rate percentile category will be derived based on the National Health Statistical Reports on resting pulse rate reference data for children, adolescents, and adults: United States, 1999-2008 (Ostchega et al. 2011). See Appendix 7 for details in deriving heart rate percentile category adjusting for age and gender.

#### 5.9 Events to Monitor

The definition for each type of adverse events to monitor is as follows:

- Injection Site Reaction is defined by preferred terms under the Medical Dictionary for Regulatory Activities (MedDRA) high-level term (HLT) "Injection site reaction".
- Immunogenicity AE: Defined using relevant PTs in the narrow SMQs for "Hypersensitivity".
- Hyperphosphatemia AE: Defined by using PTs: "Hyperphosphataemia", "Blood phosphorus increased", "Blood phosphorus abnormal".
- Ectopic calcification related AE: There is no available SMQ. Ectopic calcification related AE is defined using a MedDRA search of 'calcification'.
- Restless leg syndrome AE: Defined by PTs "Restless legs syndrome", "Restlessness", "Akathisia", "Sensory disturbance", "Psychomotor hyperactivity", "Limb discomfort", "Neuromuscular pain", "Formication".

Please see the search criteria in Appendix 8 for more details.




# 5.10 Dose Limiting Toxicity

A DLT is defined as the occurrence of any of the following:

- Unexpected SAEs occurring during treatment considered to be either definitely, probably, or possibly related to the investigational product
- A confirmed serum phosphorus level of  $\geq 6.5$  mg/dL (defined as hyperphosphatemia) at any time after dosing

If a subject experiences a DLT, the planned dosing for that subject will be evaluated by the Investigator and medical monitor. The outcome of this investigation will determine the subjects' continuation or withdrawal from the study.

#### 5.11 Duration of SOC

The definition for duration of SOC is as the following:

Duration of SOC = End date of the last SOC taken - start date of first SOC taken + 1 day

If the date is partially or completely missing, apply the following imputation rule:

#### Start Dates

- If the FIRST start date of SOC is completely missing, then use the next earliest non-missing date.
- If the year is known and month is missing, then assign 'January 1st';
- If the year and month are both known and day is missing, then assign the first day of the month.

## Stop Dates

- If LAST stop date is completely missing, then impute 'one day' prior to the inform consent date
- If year is known the month is missing, then assign "December 31<sup>st</sup>". If this imputed date is after the informed consent date, use one day prior to the informed consent date instead.

If year and month are both known and the day is missing, then assign the last day of the month. If this imputed date is after the informed consent date, use one day prior to the informed consent date instead




# **6 ANALYSIS POPULATIONS**

# 6.1 Efficacy Analysis Set

The Efficacy Analysis population will consist of all subjects who receive at least one dose of study drug and have at least one post-study drug measurement of serum phosphorus.

# 6.2 Safety Analysis Set

The Safety Analysis Set will consist of all subjects who receive at least one dose of study drug.

# 6.3 Pharmacokinetic (PK) and Pharmacodynamic (PD) Analysis Set

The PK/PD analyses sets will consist of all subjects who receive at least one dose of study drug and have evaluable blood samples.




#### 7 DATA SCREENING AND ACCEPTANCE

# 7.1 General Principles

Data will be reviewed periodically. Any questionable data will be reported to clinical data manager promptly for query and resolution.

## 7.2 Handling of Missing and Incomplete Data

Missing clinical outcome data can occur for multiple reasons, including missed subject visits and scales or measures with missing item scores. Missing and incomplete data will be identified through a review of tables and listings for this study. Missing and incomplete data will be identified for investigation, and possible resolution, by Data Management prior to the study database lock or database snapshot.

If not specified, only the actual data (not imputed data) will be presented in listings.

## 7.2.1 Missing Date Information for Adverse Events and Concomitant Medications

The following conventions will be used to impute missing portions of dates for adverse events and concomitant medications. Note that the imputed values outlined here may not always provide the most conservative date.

# Missing Start Dates

- If the day is unknown, then:
  - o If the month and year match the first dose of investigational product start date month and year in this study, then impute the day of the first dose date.
  - Otherwise, assign the first day of the month.
- If the month is unknown, then:
  - o If the year matches the year of the first dose of investigational product date in this study, then impute the month and day of the first dose date in this study.
  - Otherwise, assign 'January'
- If the year is unknown, then the date will not be imputed and will be assigned a missing value.
- If the imputed date is earlier than birth date, then birth date will be used.

#### Missing Stop Dates for events not ongoing

- If the day is unknown, then assign the last day of the month.
- If the month is unknown, then assign 'December.'
- If the year is unknown, then the date will not be imputed and will be assigned a missing value, and the event will be considered ongoing. If the AE has been recorded




as resolved/recovered, all efforts should be made to obtain the date from the Investigator.

• If the resulting end date is after the date of study completion / discontinuation/ data cutoff, set the imputed end date as the date of study completion / discontinuation/ data cutoff.

If the year is missing for the start date, and stop date (observed or imputed) is on or after the first dose or event is ongoing. The start date will be imputed as the first dose date.

# 7.2.2 Missing Causal Relationship to Investigational Product for Adverse Events

If the causal relationship to the investigational product is missing for an AE that started on or after the date of the first dose of investigational product, a causality of "definitely related" will be assigned. The imputed values for causal relationship to investigational product will be used for the incidence summary; the values will be shown as missing in the data listings.

## 7.3 Unscheduled and Early Termination Visits

Unscheduled visit occurred prior to or on the date of initiation of the first dose will be mapped to the baseline visit if it is the last assessment prior to or on the date of initiation of the first dose; otherwise no mapping will be performed.

Unscheduled visits that occurred after the date of initiation of the first dose will be mapped to the post-baseline scheduled visit with the closet target study day (refer to Section 5.2 for study day definition and Appendix 3 for the schedule of events). If the unscheduled visit is in the middle of two scheduled visits, map to the later scheduled visit.

For descriptive summary tables, when more than one measurement is mapped to the same scheduled visit, the measurement taken on the scheduled visit will be used if it is not missing, otherwise the one closest to the target day will be used. If two or more visits have equal distances to the target day, then the later one will be used. If more than one measurement is collected on the same day, use the time or the sequence number to select the latest record.

For listings and shift tables, all data points will be included.

Early termination visit will generally follow the same rule as unscheduled visit except for a special case in X-rays. X-rays will not be performed at the early termination visit if the assessment was conducted within 3 months of termination. Hence if a subject has X-rays at both Week 40 and early termination visits, the X-rays on early termination visit will be mapped to Week 64.

## 7.4 Software

SAS<sup>®</sup> software version 9.4 or higher will be used to perform all statistical analyses.




#### 8 STATISTICAL METHODS OF ANALYSES

## 8.1 General Principles

The efficacy analyses for PK/PD parameters will be based on PK/PD Analysis Set, other efficacy analyses (RGI-C, RSS and growth) will be based on the Efficacy Analysis Set, and safety analyses will be based on Safety Analysis Set. Descriptive statistics will be used to summarize the data. For continuous variables, the mean, standard deviation, standard error, median, interquartile range (Q1, Q3), minimum, and maximum will be provided. For discrete data, the frequency and percent distributions will be provided. Statistical tests will be two-sided at the alpha = 0.05 significance level. Two-sided 95% confidence intervals will also be presented. In general, missing data will be treated as missing and no statistical imputation method will be used unless stated otherwise. No adjustment on multiplicity will be made for statistical comparisons unless stated otherwise. All data obtained from the CRFs as well as any derived data will be included in data listings.

## 8.2 Subject Accountability

The number and percentage of subjects in each study population will be summarized. Screen-failure subjects and the associated reasons for failure to randomize will be tabulated. The number and percentage of subjects who complete the treatment period and of subjects who prematurely discontinue will be presented. The reasons for premature discontinuation from treatment period will be presented.

#### **8.3** Protocol Deviations

All protocol deviations will be presented in listings.

## 8.4 Investigational Product Administration

The total dose administered and weight-based dose will be summarized by study visit.

## 8.5 Demographic and Baseline Characteristics

The following demographic parameters and baseline characteristics will be summarized descriptively for the Efficacy Analysis Set:

- Age
- Gender
- Ethnicity
- Race
- Recumbent length/standing height
- Weight
- BMI




• SOC duration, age when SOC initiated

RSS scores

• XLH biochemical parameters

PHEX mutation

Renal ultrasound scores

#### 8.6 Prior and Concomitant Medication

Prior medication is defined as any medication started before the date of the first dose of investigational product (medication start date prior to the first dose date). Concomitant medication is defined as any medication taken on or after the date of the first dose of investigational product [medication end date on or after first dose date (or ongoing), and medication start date prior or on the last dose date]. Any concomitant medications started after the date of the last dose of investigational product will not be presented in the summary tables but will be included in the subject data listings. If start date is completely missing and end date is before first dose date, the medication will be considered as prior, otherwise it will be considered as concomitant.

Both prior and concomitant medications will be coded by drug name and therapeutic class using WHODRUG version 2015Q3 or the latest version at the time of snapshot/database lock. If a subject took a specific medication multiple times or took multiple medications within a specific therapeutic class, that subject would be counted only once for the coded drug name or therapeutic class.

## 8.7 Medical History / XLH Medical and Family History

Medical history will be coded by MedDRA version 18.1 or the latest version at the time of snapshot/database lock. Counts and percentages of subjects with medical history will be tabulated by system organ class and preferred term. Subject level listings for the pre-existing medical conditions, XLH medical history and family history will be provided.

# 8.8 Efficacy Analysis

The efficacy analyses for PD parameters will be performed on PK/PD Analysis Set. The efficacy analyses for clinical endpoints (RSS, RGI-C and growth) will be performed on Efficacy Analysis Set.

# 8.8.1 Generalized Estimating Equations Model

By-visit analyses using the Generalized Estimating Equations (GEE) model will be presented for all efficacy parameters. The GEE model will include study visit as categorical variables. To model the covariance structure, the exchangeable covariance matrix will be selected initially. If the exchangeable covariance structure leads to non-convergence, independence covariance structure will be applied. 95% confidence intervals (CIs) and p-values will be provided for statistical significance assessment. Baseline measures will be used as covariates.




For example, baseline RSS score will be used in the modeling for change in baseline in RSS score and for RGI-C score. Age and gender may also be used as covariates in growth endpoint models.

#### 8.8.2 Primary Efficacy Endpoint

The primary efficacy endpoint is the change from baseline over time in serum phosphorus. Descriptive statistics will be provided for observed value in serum phosphorus, change from baseline and percentage of change from baseline at each visit. The GEE model will be applied to obtain the 95% CIs and p-values. Baseline serum phosphorus measures may be included as covariate in the model.

The proportion of subjects achieving the normal range (3.2-6.1 mg/dL) will be reported. The percentage of time a subject reaches the normal range of serum phosphorus will also be summarized.

In addition, graphs showing the change of serum phosphorus over time will be provided.

## 8.8.3 Secondary Efficacy Endpoints

#### 8.8.3.1 RGI-C

The efficacy analyses evaluating RGI-C scores will be performed at Week 40 and Week 64. The GEE model will be applied to each RGI-C score type (wrist, knee, global and lower limb deformity) separately to obtain 95% CIs and p-values. Baseline RSS score will be included as a covariate in the model; age may also be included as covariate in the model. As sensitivity analysis, t test will be performed for RGI-C scores at Week 40 and Week 64. In the case when model assumption is not met, analyses using alternative methods such as non-parametric tests will be performed.

Descriptive statistics for all RGI-C scores will be provided in both continuous and categorical summary. RGI-C responder rate will be calculated. Summary of abnormality at baseline and change in abnormality at Week 40 and Week 64 will also be presented.

#### 8.8.3.2 RSS

The efficacy analyses evaluating change from Baseline of RSS scores will be performed at Week 40 and Week 64. The GEE model will be applied to each RSS score type (wrist, knee and total) separately to obtain 95% CIs and p-values. Baseline RSS score and age may be included as covariate in the model. As sensitivity analysis, t test will be performed for RSS scores at Week 40 and Week 64. In the case when the model assumption is not met, analyses using alternative methods such as non-parametric tests will be performed.

Descriptive statistics for all RSS scores and change from baseline in RSS score will be provided in both continuous and categorical summary.




#### 8.8.3.3 Growth

Growth in standing height/recumbent length and weight will be summarized over time in observed value, Z-score and percentile. Individual subject growth curves will be plotted with CDC growth charts as reference. Historical growth records may be used to evaluate change in growth velocity from pre- to post-baseline.

For standing height/recumbent length Z-score, the GEE model will be applied to obtain 95% CIs and p-values on all scheduled visits. Baseline Z score, age and gender may be included as covariate in the model.

## 8.8.4 Other Pharmacodynamics Parameters

Other PD parameters such as ALP, 1,25(OH)<sub>2</sub>D and urine phosphorus will be summarized descriptively. Summary statistics will be provided for observed value, change from baseline and percentage of change from baseline at each visit. Graphic display will be provided to show the change in PD parameters over time.

#### 8.9 Pharmacokinetics

The PK analysis will be performed on the PK/PD Analysis Set, unless stated otherwise. The descriptive statistics for serum KRN23 will be tabulated. The listing of serum KRN23 will also be provided.

The PK modeling will be detailed in a separate PK analysis plan.

#### 8.10 Safety Analysis

The safety analysis will be performed using the Safety Analysis Set. The safety parameters will include adverse events (AEs) and clinical laboratory, vital sign, physical examination, renal ultrasounds, and electrocardiographic (ECG) parameters.

#### 8.10.1 Adverse Events

Adverse events will be coded by system organ class and preferred term using the MedDRA version 18.1 or the latest version at the time of snapshot/database lock. An AE (classified by preferred term) will be considered as a treatment emergent adverse event (TEAE) if it occurred on or after the first dose and was not present prior to the first dose, or it was present at the first dose but increased in severity during the study.

An overall summary table of AEs will be presented that will summarize the frequency and percentage of subjects who experienced any AE, events to monitor, experienced any TEAE, experienced a treatment-related TEAE, a treatment-emergent SAE, discontinued from study or from study drug treatment due to a TEAE, and experienced an AE leading to death. For this purpose, a treatment-related AE is defined as an AE that is either definitely, possibly or probably related to study medication.




Subject incidence of TEAEs will be tabulated in the following manner: by system organ class/preferred term, by system organ class/preferred term/relationship to study drug, by system organ class/preferred term/severity, and by preferred term for each event to monitor category. In addition, treatment-emergent SAEs, TEAEs leading to study discontinuations and TEAEs leading to death will be tabulated by system organ class/preferred term.

The incidence of injection site reactions will be summarized by study period to assess the trend over time. The summary of incidence over time may also be explored for other events to monitor categories.

Listings will be created for AEs which lead to death, discontinuation of treatment, and SAEs.

#### 8.10.2 Safety Lab Parameters

Clinical laboratory data will be summarized by the type of laboratory test. Descriptive statistics will be calculated for each laboratory analyte at baseline and at each scheduled time point. Shift table for iPTH at each scheduled visit will be provided to assess to the normality over time. The frequency and percentage of subjects who experience abnormal clinical laboratory results and/or clinically significant abnormalities will be presented for each clinical laboratory measurement.

## 8.10.3 Physical Examination

Physical exam results will include the assessment of general appearance; head, eyes, ears, nose, and throat (HEENT); the cardiovascular, dermatology, lymphatic, respiratory, gastrointestinal, genitourinary, musculoskeletal, and neurological systems. The number and percentage of subjects with Normal/Abnormal assessment for each body system will be summarized by visit. All physical examination assessments will be listed.

#### 8.10.4 Vital Signs

Blood pressure measurements will be obtained only in children aged 3 and 4 years of age and will only be obtained at clinic visits. The blood pressure will be summarized by study visit in mmHg and percentile to assess the blood pressure change over time. The average of the triple measurements will be used in the summary.

Heart rate and heart rate percentile category will also be summarized by study visit.

## 8.10.5 Renal Ultrasound

Renal ultrasound will be conducted with findings of nephrocalcinosis graded on a 5-point scale by a central reader. The renal ultrasound is read using a pre-defined methodology (Biomedical Systems Independent Review Manual November 2014). These results will be summarized by time point, a grade shift table summarizing changes from Baseline by time point will also be created.




# 8.10.6 Electrocardiogram

Descriptive statistics for ECG parameters (heart rate, RR interval, PR interval, QRS duration, QT interval, and QTc) and changes from baseline values at each assessment time point to the end of study will be presented by. The QTc will be calculated using both the Bazett and Fridericia corrections.

ECG parameters will be summarized by the maximum post-baseline value and maximum change from baseline using the following categories based on FDA guidance (FDA 2015) listed in Table 8.10.6.1.

**Table 8.10.6.1:** Criteria for ECG Results

| ECG Parameter | Categories for Baseline and<br>Maximum Post-Baseline Value | Categories for Maximum Change<br>from Baseline Value |
|---|---|---|
| PR Interval | ≤200 and >200 msec | ≤20 and >20 msec |
| QRS Interval | ≤110 and >110 msec | ≤10 and >10 msec |
| QTc Interval | ≤450, >450-≤480, >480-≤500 and >500 msec | ≤30, >30-≤60 and >60 msec |




## 9 REFERENCES

- Biomedical Systems Independent Review Manual July. 2015. "Independent review manual of X-ray RGI-C for UX023-CL201 study, dated July 21, 2015."
- Biomedical Systems Independent Review Manual November. 2014. "Independent review manual of Ultrasound for UX023-CL201 study, dated November 14, 2014."
- Biomedical Systems Independent Review Manual September. 2014. "Independent review manual of X-ray RSS for UX023-CL201 study, dated September 29, 2014."
- Kuczmarski, RJ, Ogden, CL, Grummer-Strawn, LM, Flegal, KM, Guo, SS, Wei, R, Mei, Z, Curtin, LR, Roche, AF, and Johnson, CL. 2000. "CDC growth charts: United States." *Adv Data* (314):1-27.
- NHLBI. 2005. "The Fourth Report on the Diagnosis, Evaluation, and Treatment of High Blood Pressure in Children and Adolescents. National Institutes of Health." *National Heart, Lung, and Blood Institute*.
- Ostchega, Y, Porter, KS, Hughes, J, Dillon, CF, and Nwankwo, T. 2011. "Resting pulse rate reference data for children, adolescents, and adults: United States, 1999-2008." *Natl Health Stat Report* (41):1-16.
- Thacher, TD, Fischer, PR, Pettifor, JM, Lawson, JO, Manaster, BJ, and Reading, JC. 2000. "Radiographic scoring method for the assessment of the severity of nutritional rickets." *J Trop Pediatr* 46 (3):132-9.




# 10 APPENDICES

# **Appendix 1: Efficacy Endpoint Summary Table**

| | | Analysis | | Data Time | | Week 64 |
|---|---|---|---|---|---|---|
| Endpoints | Scale | Set | Comparisons | Points | Week 40 Analysis | Analysis |
| Serum phosphorus | Continuous | PK/PD | Baseline vs. | Refer to | GEE | GEE |
| | | | Post-baseline | Schedule of | Descriptive | Descriptive |
| | | | | Events | Statistics | Statistics |
| | | | | (Appendix 3) | | |
| RGI-C wrist, knee, | Continuous | Efficacy | Baseline vs. | Baseline, | GEE | GEE |
| global and lower limb | Categorical | | Post-baseline | Week 40, 64 | Descriptive | Descriptive |
| deformity scores | | | | | Statistics | Statistics |
| RSS knee, wrist and total | Continuous | Efficacy | Baseline vs. | Baseline, | GEE | GEE |
| scores | | | Post-baseline | Week 40, 64 | Descriptive | Descriptive |
| | | | | | Statistics | Statistics |
| Growth (standing | Continuous | Efficacy | Baseline vs. | Baseline, | GEE | GEE |
| height/recumbent length) | | | Post-baseline | Week 12, 24, | Descriptive | Descriptive |
| | | | | 40, 64 | Statistics | Statistics |
| Other PD parameters | Continuous | PK/PD | Baseline vs. | Refer to | Descriptive | Descriptive |
| F | | | Post-baseline | Schedule of | Statistics | Statistics |
| | | | | Events | | |
| | | | | (Appendix 3) | | |
| | | | | (TPP CHAIN 3) | | |
| Ĺ | 1 | _1 | | I | | 1 |

Page 28 Proprietary and Confidential




# **Appendix 2: Clinical Laboratory Assessments for Safety**

| Chemistry | Hematology | Urinalysis <sup>1</sup> |
|---|---|---|
| $1,25(OH)_2D^2$ | Hematocrit | Appearance |
| 25(OH) <sub>2</sub> D | Hemoglobin | Color |
| Alanine aminotransferase (ALT) | Platelet count | pH |
| Alkaline phosphatase (ALP) <sup>2</sup> | Red blood cell (RBC) count | Specific gravity |
| Amylase | White blood cell (WBC) count | Ketones |
| Aspartate aminotransferase (AST) | Mean corpuscular volume (MCV) | Protein |
| Bilirubin (direct and total) | Mean corpuscular hemoglobin (MCH) | Glucose |
| Blood urea nitrogen (BUN) | MCH concentration | |
| Calcium (total) | | |
| Chloride | | |
| Carbon dioxide (CO <sub>2</sub> ) | | |
| Cholesterol (total) | | |
| Creatinine | | |
| Gamma-glutamyl transpeptidase (GGT) | | |
| Glucose | | |
| FGF23 | | |
| Intact parathyroid hormone (iPTH) | | |
| Lactate dehydrogenase (LDH) | | Spot Urine |
| Lipase | | Calcium |
| Phosphorus <sup>2</sup> | | Creatinine |

Page 29 Proprietary and Confidential




| Chemistry | Hematology | Urinalysis <sup>1</sup> |
|-----------------------------|------------|-------------------------|
| Potassium | | Phosphorus |
| Protein (albumin and total) | | |
| Sodium | | |
| Uric acid | | |

<sup>&</sup>lt;sup>1</sup>Urinalysis to be conducted if possible based on urine volume collected. <sup>2</sup>Also designated as a PD/efficacy parameter

Statistical Analysis Plan




# Appendix 3: Schedule of Events

Table 10.1: Schedule of Events – Screening, Baseline, and Treatment Period Weeks 1-30

| | Screen<br>Baseli | ing/<br>ine <sup>1</sup> | | | | | | | | Treat | ment l | Period <sup>3</sup> | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| VISIT TYPE/NUMBER | sv | BL<br>V1 <sup>2</sup> | HH <sup>4</sup><br>V2 | HH<br>V3 | V4 | HH<br>V5 | V6 | HH<br>V7 | V8 | HH<br>V9 | V10 | HH<br>V11 | HH<br>V12 | V13 | HH<br>V14 | V15 | HH<br>V16 | HH<br>V17 | HH<br>V18 |
| WEEK | W -6<br>to BL | W0 | W1 | W2 | W4 | W6 | W8 | W<br>10 | W<br>12 | W<br>14 | W<br>15 | W<br>16 | W<br>18 | W<br>20 | W<br>22 | W<br>24 | W<br>26 | W<br>28 | W<br>30 |
| Informed Consent | X | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | X | X | | | | | | | | | | | | | | | | | |
| Medical History &<br>Demographics | X | | | | | | | | | | | | | | | | | | |
| PHEX mutation analysis 5 | X | | | | | | | | | | | | | | | | | | |
| PD MEASURES | | | | | | | | | | | | | | | | | | | |
| Serum Phosphorus <sup>6</sup> | | X | X | | X | | X | | X | | X | | | X | | | | | |
| 1,25(OH) <sub>2</sub> D <sup>6</sup> | | X | X | | | | | | X | | | | | X | | | | | |
| Spot urine <sup>6,7</sup> | | X | | | X | | | | X | | X | | | X | | | | | |
| ALP only <sup>6</sup> | | X | | | | | | | | | | | | X | | | | | |
| EFFICACY MEASURES | | | | | | | | | | | | | | | | | | | |
| Growth (recumbent length/standing height) | | X | | | | | | | X | | | | | | | X | | | |
| Bilateral AP knee X-rays <sup>2</sup> | X | | | | | | | | | | | | | | | | | | |
| Bilateral PA hand/wrist <sup>2</sup> | | X | | | | | | | | | | | | | | | | | |
| Standing long leg X-Ray <sup>2</sup> | | X | | | | | | | | | | | | | | | | | |
| PHARMACOKINETICS | | | | | | | | | | | | | | | | | | | |
| Serum Pre-Dose KRN23 <sup>6</sup> | | | X | | X | | | | X | | | | | | | | | | |

Proprietary and Confidential Page 31




| | Screen<br>Baseli | | | | V4 V5 V6 V7 V8 V9 V10 V11 V12 V13 V14 V15 V16 V17 V13 V4 W6 W8 W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W W < | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| VISIT TYPE/NUMBER | sv | BL<br>V1 <sup>2</sup> | HH <sup>4</sup><br>V2 | HH<br>V3 | V4 | | V6 | l | V8 | | V10 | | | V13 | l | V15 | | | HH<br>V18 |
| WEEK | W -6<br>to BL | W0 | W1 | W2 | W4 | W6 | W8 | | | | | | | | | | | | W<br>30 |
| SAFETY | | | | | | | | | | | | | | | | | | | |
| Vital Signs 8,9 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Weight | X | X | | | X | | | | X | | | | | | | X | | | |
| Physical Examination | X | X | | | | | | | | | | | | | | X | | | |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Renal Ultrasound <sup>2</sup> | X | | | | | | | | | | | | | | | | | | |
| ECG <sup>2</sup> | | X | | | | | | | X | | | | | | | | | | |
| Chemistry, Hematology,<br>Urinalysis <sup>6,7,10</sup> | X | X | | | X | | | | X | | | | | X | | | | | |
| Serum 25(OH)D <sup>6</sup> | X | | | | | | | | X | | | | | | | | | | |
| Serum Calcium <sup>6</sup> | X | X | X | | X | | X | | X | | X | | | X | | | | | |
| Serum Creatinine <sup>6</sup> | X | X | | | X | | | | X | | X | | | X | | | | | |
| Serum iPTH <sup>6</sup> | X | X | | | | | | | X | | | | | X | | | | | |
| Serum FGF23 <sup>6</sup> | | X | | | | | | | | | | | | | | X | | | |
| Anti-KRN23 antibody<br>(HAHA) <sup>6,11</sup> | | X | | | X | | | | X | | | | | | | | | | |
| DRUG ADMINISTRATION | | X | | X | X | X | X | X | X | X | | X | X | X | X | X | X | X | X |

See footnotes after Table 10.2




Table 10.2: Schedule of Events – Treatment Period Weeks 32 – 64

| | | Treatment Period <sup>3</sup> | | | | | | | | | | | | | | Safety<br>Visit <sup>13</sup> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Type/Number | V19 | HH<br>V20 | HH<br>V21 | HH<br>V22 | V23 | HH<br>V24 | HH<br>V25 | HH<br>V26 | V27 | HH<br>V28 | HH<br>V29 | HH<br>V30 | V31 | HH<br>V32 | HH<br>V33 | HH<br>V34 | V35 | V36 |
| Week | W<br>32 | W<br>34 | W<br>36 | W<br>38 | W<br>40 | W<br>42 | W<br>44 | W<br>46 | W<br>48 | W<br>50 | W<br>52 | W<br>54 | W<br>56 | W<br>58 | W<br>60 | W<br>62 | W64/<br>ET <sup>12</sup> | W<br>76 |
| PD MEASURES | | | | | | | | | | | | | | | | | | |
| Serum Phosphorus <sup>6</sup> | X | | | | X | | | | X | | | | X | | | | X | X |
| 1,25(OH) <sub>2</sub> D <sup>6</sup> | X | | | | X | | | | X | | | | X | | | | X | X |
| Spot urine <sup>6,7</sup> | X | | | | X | | | | X | | | | X | | | | X | X |
| ALP only <sup>6</sup> | | | | | X | | | | | | | | | | | | X | |
| EFFICACY MEASURES | | | | | | | | | | | | | | | | | | |
| Growth (length/standing height) | | | | | X | | | | | | | | | | | | X | |
| Bilateral AP knee X-rays <sup>2</sup> | | | | | X | | | | | | | | | | | | X | |
| Bilateral PA hand/wrist<br>X-rays <sup>2</sup> | | | | | X | | | | | | | | | | | | X | |
| Standing long leg X-ray <sup>2</sup> | | | | | X | | | | | | | | | | | | X | |
| PHARMACOKINETICS | | | | | | | | | | | | | | | | | | |
| Serum Pre-Dose KRN23 <sup>6</sup> | | | | | X | | | | | | | | | | | | | |
| SAFETY | | | | | | | | | | | | | | | | | | |
| Vital Signs 8,9 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Weight | X | | | | X | | | | X | | | | X | | | | | |
| Physical Examination | | | | | X | | | | | | | | | | | | X | X |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

Statistical Analysis Plan




| | Treatment Period <sup>3</sup> | | | | | | | | | | | | | | | | Safety<br>Visit <sup>13</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Type/Number | V19 | HH<br>V20 | HH<br>V21 | HH<br>V22 | V23 | HH<br>V24 | HH<br>V25 | HH<br>V26 | V27 | HH<br>V28 | HH<br>V29 | HH<br>V30 | V31 | HH<br>V32 | HH<br>V33 | HH<br>V34 | V35 | V36 |
| Week | W<br>32 | W<br>34 | W<br>36 | W<br>38 | W<br>40 | W<br>42 | W<br>44 | W<br>46 | W<br>48 | W<br>50 | W<br>52 | W<br>54 | W<br>56 | W<br>58 | W<br>60 | W<br>62 | W64/<br>ET <sup>12</sup> | W<br>76 |
| Renal Ultrasound <sup>2</sup> | | | | | X | | | | | | | | | | | | X | |
| ECG <sup>2</sup> | | | | | X | | | | | | | | | | | | X | |
| Chemistry, Hematology,<br>Urinalysis <sup>6,7,10</sup> | | | | | X | | | | X | | | | X | | | | X | X |
| Serum 25(OH)D <sup>6</sup> | | | | | X | | | | | | | | | | | | X | |
| Serum Calcium <sup>6</sup> | X | | | | X | | | | X | | | | X | | | | X | X |
| Serum Creatinine <sup>6</sup> | X | | | | X | | | | X | | | | X | | | | X | |
| Serum iPTH <sup>6</sup> | | | | | X | | | | | | | | | | | | X | |
| Serum FGF23 <sup>6</sup> | | | | | | | | | | | | | | | | | X | |
| Anti-KRN23 antibody<br>(HAHA) <sup>6, 11</sup> | | | | | X | | | | | | | | | | | | | |
| DRUG ADMINISTRATION | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |

The baseline visit may occur up to approximately 6 weeks after Screening in those subjects without a previously documented *PHEX* mutation to allow for *PHEX* mutation results to be determined

All Screening/Baseline assessments and inclusion/exclusion criteria based on local lab results must be satisfied prior to randomization and dosing. Renal ultrasound, ECG, and x-rays may be performed within ± 3 days of clinic visit to accommodate scheduling availability.

Subjects will return to the clinic for site visits at approximately 4-week intervals from Baseline to Week 24 and at 8-week intervals from Week 24 to Week 64. The visit window is ± 3 days

Home health (HH) visits may also be conducted at the clinic depending on proximity of the subject to the investigational site and local availability of home health care resources. The visit window is ± 3 days.

PHEX mutation analysis will be performed for all subjects. Potential subjects with prior confirmation of a PHEX mutation or variant of uncertain significance in either self or a family member with appropriate X-linked inheritance who meet other eligibility requirements may enroll before screening PHEX mutation results are returned.

Statistical Analysis Plan




- Blood and urine to be collected after a minimum fasting time of 4 hours and prior to drug administration (if applicable). Record fasting duration on CRF. Subjects who live more than 45 minutes from the site may stay overnight on the night before the site visit to facilitate fasting sample collection. At Baseline, local lab values will be used to confirm eligibility. Baseline samples will also be sent to the central lab for data analysis. Serum phosphorus may be collected as an unscheduled lab if necessary
- <sup>7</sup> Spot urine collections for urinary calcium, phosphorus, and creatinine
- At site visits, vital sign measurements consist of seated systolic/diastolic blood pressure (BP) measured in millimeters of mercury (mm Hg), heart rate (HR; beats per minute), respiration rate (breaths per minute), and temperature in degrees Celsius (°C). Blood pressure will only be obtained for subjects age 3 or 4 years. Obtain HR, respiration rate, and temperature at the beginning of each visit before any additional assessments are completed. At the Screening Visit BP should be measured 3 times, 30 seconds apart at the beginning of each visit; 3 additional BP measurements, 30 seconds apart, should be obtained at the end of the study visit after all procedures have been performed. At baseline and post-baseline visits, 3 BP measurements 30 seconds apart, should be obtained at the beginning of the study visit.
- At HH visits, vital sign measurements consist of HR (beats per minute) and temperature in degrees Celsius (°C). Obtain at the beginning of each visit before any additional assessments are completed.
- Serum chemistry panels may include PD parameters (i.e., serum phosphorus and ALP), and safety parameters of interest (i.e., calcium) to avoid duplication of testing. Urinalysis will be conducted if possible based on urine volume collected.
- 11 If the development of anti-KRN23 antibodies is suspected in a given subject, samples may be obtained at additional time points on a case-by-case basis, if warranted.
- Radiography (x-rays) will not be performed at the early termination (ET) visit if the assessment was conducted within 3 months of termination.
- An additional safety visit will take place 12 weeks ±1 week after the date of the last study drug administration for those subjects who discontinue treatment, or 12 weeks ±1 week after the Week 64 visit for subjects who complete the study and choose not to enroll immediately in an extension study. This visit is not required for subjects who are eligible and choose to take part in an extension study. Every reasonable effort should be made to have required subjects return to the clinic for the final safety visit; however, subjects who are unable to return to the clinic for the final safety visit will be given the option of providing blood and urine samples as part of a HH visit.

Statistical Analysis Plan




# **Appendix 4: RSS Data Collection Form**

# **WRIST**

| GR | GRADE DEFINITIONS FOR RADIUS AND ULNA based on radiographic features below | |
|---|---|---|
| | 1 | Widened growth plate, irregularity of metaphyseal margin, but without concave cupping |
| | 2 | Metaphyseal concavity with fraying of margins |




Statistical Analysis Plan




# **KNEE**

| GRADE DEFIN | ITIONS FOR FEMUR AND TIBIA based on the degree of lucency and widening of zone of provisional calcification |
|---|---|
| 1 | Partial lucency, smooth margin of metaphysis visible |
| 2 | Partial lucency, smooth margin of metaphysis NOT visible |
| 3 | Complete lucency, epiphysis appears widely separated from distal metaphysis |

| Grade femur<br>circle 1, 2, or 3 | FEMUR | 2 3 | Determine multiplier for femur circle 0.5 or 1 Based on portion of growth plate affect ≤ one condyle or plateau affected Two condyles or plateaus affected | 0.5<br>1 |
|---|---|---|---|---|
| Grade tibia<br>circle 1, 2, or 3 | TIBIA | 2 3 | Determine multiplier for tibia circle 0.5 or 1 Based on portion of growth plate affected ≤ one condyle or plateau affected Two condyles or plateaus affected | 0.5 |



Version 15Aug2010

Proprietary and Confidential Page 37

Statistical Analysis Plan




# **Appendix 5: RGI-C Data Collection Form**

### REGIONAL RATING OF RICKETS

How would you rate the change in XLH-related rickets in the HANDS/WRISTS? Circle one

| -3 | -2 | -1 | 0 | +1 | +2 | +3 |
|---|---|---|---|---|---|---|
| Severe<br>Worsening | Moderate<br>Worsening | Minimal<br>Worsening | No Change | Minimal<br>Healing | Substanti al<br>Healing | Complete or Near<br>Complete Healing |

Identify abnormalities in image A on the left and then rate any change seen in image B on the right compared to image A

#### PA HAND/WRIST SINGLE ABNORMALITY RATING **BILATERAL PA RADIUS** NOT in "A" DECREASED | UNCHANGED | INCREASED Metaphyseal lucency Metaphyseal/epiphyseal separation Metaphyseal fraying Metaphyseal concavity **BILATERAL PA ULNA** DECREASED NOT in "A" UNCHANGED INCREASED Metaphyseal lucency Metaphyseal/epiphyseal separation Metaphyseal fraying Metaphyseal concavity

Statistical Analysis Plan




## REGIONAL RATING OF RICKETS

How would you rate the change in XLH-related rickets in the KNEES? Circle one

| -3 | -2 | -1 | 0 | +1 | +2 | +3 |
|---|---|---|---|---|---|---|
| Severe<br>Worsening | Moderate<br>Worsening | Minimal<br>Worsening | No Change | Minimal<br>Healing | Substanti al<br>Healing | Complete or Near<br>Complete Healing |

Identify abnormalities in image A on the left and then rate any change seen in image B on the right compared to image A

## AP KNEES SINGLE ABNORMALITY RATING

| BILATERAL AP FEMUR | NOT in "A" | DECREASED | UNCHAN GED | INCREASED |
|---|---|---|---|---|
| Metaphyseal lucency | | | | |
| Metaphyseal/epiphyseal separation | | | | |
| Metaphyseal fraying | | | | |
| Metaphyseal concavity | | | | |

Statistical Analysis Plan




## AP KNEES SINGLE ABNORMALITY RATING

| BILATERAL AP TIBIA | NOT in "A" | DECREASED | UNCHAN GED | INCREASED |
|---|---|---|---|---|
| Metaphyseal lucency | | | | |
| Metaphyseal/epiphyseal separation | | О | | |
| Metaphyseal fraying | | | | |
| Metaphyseal concavity | | | | |
| BILATERAL AP FIBULA | NOT in "A" | DECREASED | UNCHAN GED | INCREASED |
| BILATERAL AP FIBULA Metaphyseal lucency | | DECREASED | UNCHAN GED | INCREASED |
| Metaphyseal lucency | | | | |

Statistical Analysis Plan




## **GLOBAL RATING OF RICKETS**

How would you rate the change in XLH-related rickets?

The B images on the right as compared to A images on the left show circle one

| -3 | -2 | -1 | 0 | +1 | +2 | +3 |
|---|---|---|---|---|---|---|
| Severe<br>Worsening | Moderate<br>Worsening | Minimal<br>Worsening | No Change | Minimal<br>Healing | Substantial<br>Healing | Complete or<br>Near Complete<br>Healing |

### RATING OF LOWER LIMB DEFORMITY

How would you rate the change in XLH-related lower limb deformity? Circle one

| -3 | -2 | -1 | 0 | +1 | +2 | +3 |
|---|---|---|---|---|---|---|
| Severe<br>Worsening | Moderate<br>Worsening | Minimal<br>Worsening | No Change | Minimal<br>Healing | Substanti al<br>Healing | Complete or Near<br>Complete Healing |

Identify abnormalities in image A on the left and then rate any change seen in image B on the right compared to image A

## SINGLE ABNORMALITY RATING

| STANDING LONG LEG | NOT in "A" | VARUS | VALGUS | DECREASED | UNCHAN GED | INCREASED |
|---|---|---|---|---|---|---|
| L Tibia | | | | | | |
| R Tibia | | | | | | |
| L Fibula | | | | | | |
| R Fibula | | | | | | |
| L Femur | | | | | | |
| R Femur | | | | | | |



Appendix 6: Blood Pressure Percentiles by Gender, Age and Height (NHLBI 2005)









**Appendix 7: Heart Rate Percentiles by Gender and Age** 






# **Appendix 8: Events to Monitor**

Injection site reactions: based on HLT "Injection site reaction"

| Category | PT |
|-------------------------|----------------------------------|
| Injection site reaction | Embolia cutis medicamentosa |
| Injection site reaction | Injected limb mobility decreased |
| Injection site reaction | Injection site abscess |
| Injection site reaction | Injection site abscess sterile |
| Injection site reaction | Injection site anaesthesia |
| Injection site reaction | Injection site atrophy |
| Injection site reaction | Injection site bruising |
| Injection site reaction | Injection site calcification |
| Injection site reaction | Injection site cellulitis |
| Injection site reaction | Injection site coldness |
| Injection site reaction | Injection site cyst |
| Injection site reaction | Injection site dermatitis |
| Injection site reaction | Injection site discharge |
| Injection site reaction | Injection site discolouration |
| Injection site reaction | Injection site discomfort |
| Injection site reaction | Injection site dryness |
| Injection site reaction | Injection site dysaesthesia |
| Injection site reaction | Injection site eczema |
| Injection site reaction | Injection site erosion |
| Injection site reaction | Injection site erythema |
| Injection site reaction | Injection site exfoliation |
| Injection site reaction | Injection site extravasation |
| Injection site reaction | Injection site fibrosis |
| Injection site reaction | Injection site granuloma |
| Injection site reaction | Injection site haematoma |
| Injection site reaction | Injection site haemorrhage |
| Injection site reaction | Injection site hyperaesthesia |
| Injection site reaction | Injection site hypersensitivity |
| Injection site reaction | Injection site hypertrichosis |
| Injection site reaction | Injection site hypertrophy |
| Injection site reaction | Injection site hypoaesthesia |
| Injection site reaction | Injection site induration |
| Injection site reaction | Injection site infection |
| Injection site reaction | Injection site inflammation |
| Injection site reaction | Injection site injury |
| Injection site reaction | Injection site irritation |
| Injection site reaction | Injection site ischaemia |
| Injection site reaction | Injection site joint discomfort |



| Category | PT |
|-------------------------|------------------------------------------|
| Injection site reaction | Injection site joint effusion |
| Injection site reaction | Injection site joint erythema |
| Injection site reaction | Injection site joint infection |
| Injection site reaction | Injection site joint inflammation |
| Injection site reaction | Injection site joint movement impairment |
| Injection site reaction | Injection site joint pain |
| Injection site reaction | Injection site joint swelling |
| Injection site reaction | Injection site joint warmth |
| Injection site reaction | Injection site laceration |
| Injection site reaction | Injection site lymphadenopathy |
| Injection site reaction | Injection site macule |
| Injection site reaction | Injection site mass |
| Injection site reaction | Injection site movement impairment |
| Injection site reaction | Injection site necrosis |
| Injection site reaction | Injection site nerve damage |
| Injection site reaction | Injection site nodule |
| Injection site reaction | Injection site oedema |
| Injection site reaction | Injection site pain |
| Injection site reaction | Injection site pallor |
| Injection site reaction | Injection site papule |
| Injection site reaction | Injection site paraesthesia |
| Injection site reaction | Injection site phlebitis |
| Injection site reaction | Injection site photosensitivity reaction |
| Injection site reaction | Injection site plaque |
| Injection site reaction | Injection site pruritus |
| Injection site reaction | Injection site pustule |
| Injection site reaction | Injection site rash |
| Injection site reaction | Injection site reaction |
| Injection site reaction | Injection site recall reaction |
| Injection site reaction | Injection site scab |
| Injection site reaction | Injection site scar |
| Injection site reaction | Injection site streaking |
| Injection site reaction | Injection site swelling |
| Injection site reaction | Injection site thrombosis |
| Injection site reaction | Injection site ulcer |
| Injection site reaction | Injection site urticarial |
| Injection site reaction | Injection site vasculitis |
| Injection site reaction | Injection site vesicles |
| Injection site reaction | Injection site warmth |
| Injection site reaction | Malabsorption from injection site |




Immunogenicity: based on relevant PTs in the narrow SMQs for "Hypersensitivity"

| Category | PT |
|------------------|----------------------------------------------------------|
| Hypersensitivity | Acute generalised exanthematous pustulosis |
| Hypersensitivity | Administration site dermatitis |
| Hypersensitivity | Administration site eczema |
| Hypersensitivity | Administration site hypersensitivity |
| Hypersensitivity | Administration site rash |
| Hypersensitivity | Administration site recall reaction |
| Hypersensitivity | Administration site urticaria |
| Hypersensitivity | Administration site vasculitis |
| Hypersensitivity | Allergic bronchitis |
| Hypersensitivity | Allergic colitis |
| Hypersensitivity | Allergic cough |
| Hypersensitivity | Allergic cystitis |
| Hypersensitivity | Allergic eosinophilia |
| Hypersensitivity | Allergic gastroenteritis |
| Hypersensitivity | Allergic granulomatous angiitis |
| Hypersensitivity | Allergic hepatitis |
| Hypersensitivity | Allergic keratitis |
| Hypersensitivity | Allergic myocarditis |
| Hypersensitivity | Allergic oedema |
| Hypersensitivity | Allergic otitis externa |
| Hypersensitivity | Allergic otitis media |
| Hypersensitivity | Allergic pharyngitis |
| Hypersensitivity | Allergic respiratory disease |
| Hypersensitivity | Allergic respiratory symptom |
| Hypersensitivity | Allergic sinusitis |
| Hypersensitivity | Allergic transfusion reaction |
| Hypersensitivity | Allergy alert test positive |
| Hypersensitivity | Allergy test positive |
| Hypersensitivity | Allergy to immunoglobulin therapy |
| Hypersensitivity | Allergy to vaccine |
| Hypersensitivity | Alveolitis allergic |
| Hypersensitivity | Anaphylactic reaction |
| Hypersensitivity | Anaphylactic shock |
| Hypersensitivity | Anaphylactic transfusion reaction |
| Hypersensitivity | Anaphylactoid reaction |
| Hypersensitivity | Anaphylactoid shock |
| Hypersensitivity | Anaphylaxis treatment |
| Hypersensitivity | Angioedema |
| Hypersensitivity | Antiallergic therapy |
| Hypersensitivity | Antiendomysial antibody positive |
| Hypersensitivity | Anti-neutrophil cytoplasmic antibody positive vasculitis |
| Hypersensitivity | Application site dermatitis |
| Hypersensitivity | Application site eczema |
| Hypersensitivity | Application site hypersensitivity |

Protocol Number: UX023-CL205 Statistical Analysis Plan 29 November 2016, Version 1.0





| Category | PT |
|------------------|-------------------------------------------------------|
| Hypersensitivity | Application site rash |
| Hypersensitivity | Application site recall reaction |
| Hypersensitivity | Application site urticaria |
| Hypersensitivity | Application site vasculitis |
| Hypersensitivity | Arthritis allergic |
| Hypersensitivity | Atopy |
| Hypersensitivity | Blepharitis allergic |
| Hypersensitivity | Blood immunoglobulin E abnormal |
| Hypersensitivity | Blood immunoglobulin E increased |
| Hypersensitivity | Bromoderma |
| Hypersensitivity | Bronchospasm |
| Hypersensitivity | Catheter site dermatitis |
| Hypersensitivity | Catheter site eczema |
| Hypersensitivity | Catheter site hypersensitivity |
| Hypersensitivity | Catheter site rash |
| Hypersensitivity | Catheter site urticaria |
| Hypersensitivity | Catheter site vasculitis |
| Hypersensitivity | Chronic eosinophilic rhinosinusitis |
| Hypersensitivity | Chronic hyperplastic eosinophilic sinusitis |
| Hypersensitivity | Circulatory collapse |
| Hypersensitivity | Circumoral oedema |
| Hypersensitivity | Conjunctival oedema |
| Hypersensitivity | Conjunctivitis allergic |
| Hypersensitivity | Corneal oedema |
| Hypersensitivity | Cutaneous vasculitis |
| Hypersensitivity | Dennie-Morgan fold |
| Hypersensitivity | Dermatitis |
| Hypersensitivity | Dermatitis acneiform |
| Hypersensitivity | Dermatitis allergic |
| Hypersensitivity | Dermatitis atopic |
| Hypersensitivity | Dermatitis bullous |
| Hypersensitivity | Dermatitis contact |
| Hypersensitivity | Dermatitis exfoliative |
| Hypersensitivity | Dermatitis exfoliative generalised |
| Hypersensitivity | Dermatitis herpetiformis |
| Hypersensitivity | Dermatitis infected |
| Hypersensitivity | Dermatitis psoriasiform |
| Hypersensitivity | Distributive shock |
| Hypersensitivity | Documented hypersensitivity to administered product |
| Hypersensitivity | Drug cross-reactivity |
| Hypersensitivity | Drug eruption |
| Hypersensitivity | Drug hypersensitivity |
| Hypersensitivity | Drug provocation test |
| Hypersensitivity | Drug reaction with eosinophilia and systemic symptoms |
| Hypersensitivity | Eczema |
| Hypersensitivity | Eczema infantile |



| Category | PT |
|------------------|------------------------------------|
| Hypersensitivity | Eczema nummular |
| Hypersensitivity | Eczema vaccinatum |
| Hypersensitivity | Eczema vesicular |
| Hypersensitivity | Eczema weeping |
| Hypersensitivity | Encephalitis allergic |
| Hypersensitivity | Encephalopathy allergic |
| Hypersensitivity | Epidermal necrosis |
| Hypersensitivity | Epidermolysis |
| Hypersensitivity | Epidermolysis bullosa |
| Hypersensitivity | Epiglottic oedema |
| Hypersensitivity | Erythema multiforme |
| Hypersensitivity | Erythema nodosum |
| Hypersensitivity | Exfoliative rash |
| Hypersensitivity | Eye allergy |
| Hypersensitivity | Eye oedema |
| Hypersensitivity | Eye swelling |
| Hypersensitivity | Eyelid oedema |
| Hypersensitivity | Face oedema |
| Hypersensitivity | Giant papillary conjunctivitis |
| Hypersensitivity | Gingival oedema |
| Hypersensitivity | Gingival swelling |
| Hypersensitivity | Gleich's syndrome |
| Hypersensitivity | Haemorrhagic urticaria |
| Hypersensitivity | Hand dermatitis |
| Hypersensitivity | Henoch-Schonlein purpura |
| Hypersensitivity | Henoch-Schonlein purpura nephritis |
| Hypersensitivity | Hereditary angioedema |
| Hypersensitivity | Hypersensitivity |
| Hypersensitivity | Hypersensitivity vasculitis |
| Hypersensitivity | Idiopathic urticaria |
| Hypersensitivity | Immediate post-injection reaction |
| Hypersensitivity | Immune thrombocytopenic purpura |
| Hypersensitivity | Immune tolerance induction |
| Hypersensitivity | Infusion site dermatitis |
| Hypersensitivity | Infusion site eczema |
| Hypersensitivity | Infusion site hypersensitivity |
| Hypersensitivity | Infusion site rash |
| Hypersensitivity | Infusion site recall reaction |
| Hypersensitivity | Infusion site urticaria |
| Hypersensitivity | Infusion site vasculitis |
| Hypersensitivity | Injection site dermatitis |
| Hypersensitivity | Injection site eczema |
| Hypersensitivity | Injection site hypersensitivity |
| Hypersensitivity | Injection site rash |
| Hypersensitivity | Injection site recall reaction |
| Hypersensitivity | Injection site urticaria |





| Category | PT |
|---|---|
| Hypersensitivity | Injection site vasculitis |
| Hypersensitivity | Instillation site hypersensitivity |
| Hypersensitivity | Instillation site rash |
| Hypersensitivity | Instillation site urticaria |
| Hypersensitivity | Interstitial granulomatous dermatitis |
| Hypersensitivity | Intestinal angioedema |
| Hypersensitivity | Iodine allergy |
| Hypersensitivity | Kaposi's varicelliform eruption |
| Hypersensitivity | Kounis syndrome |
| Hypersensitivity | Laryngeal oedema |
| Hypersensitivity | Laryngitis allergic |
| Hypersensitivity | Laryngospasm |
| Hypersensitivity | Laryngotracheal oedema |
| Hypersensitivity | Limbal swelling |
| Hypersensitivity | Lip oedema |
| Hypersensitivity | Lip swelling |
| Hypersensitivity | Mast cell degranulation present |
| Hypersensitivity | Mouth swelling |
| Hypersensitivity | Mucocutaneous rash |
| Hypersensitivity | Multiple allergies |
| Hypersensitivity | Nephritis allergic |
| Hypersensitivity | Nikolsky's sign |
| Hypersensitivity | Nodular rash |
| Hypersensitivity | Oculomucocutaneous syndrome |
| Hypersensitivity | Oculorespiratory syndrome |
| Hypersensitivity | Oedema mouth |
| Hypersensitivity | Oral allergy syndrome |
| Hypersensitivity | Oropharyngeal blistering |
| Hypersensitivity | Oropharyngeal spasm |
| Hypersensitivity | Oropharyngeal swelling |
| Hypersensitivity | Palatal oedema |
| Hypersensitivity | Palatal swelling |
| Hypersensitivity | Palisaded neutrophilic granulomatous dermatitis |
| Hypersensitivity | Palpable purpura |
| Hypersensitivity | Pathergy reaction |
| Hypersensitivity | Periorbital oedema |
| Hypersensitivity | Pharyngeal oedema |
| Hypersensitivity | Pruritus allergic |
| Hypersensitivity | Radioallergosorbent test positive |
| Hypersensitivity | Rash |
| Hypersensitivity | Rash erythematous |
| Hypersensitivity | Rash follicular |
| Hypersensitivity | Rash generalised |
| Hypersensitivity | Rash macular |
| | Rash maculo-papular |
| Hypersensitivity Hypersensitivity | Rash maculovesicular |
| Trypersensitivity | INASII IIIACUIOVESICUIAI |



| Category | PT |
|------------------|-------------------------------------------|
| Hypersensitivity | Rash morbilliform |
| Hypersensitivity | Rash neonatal |
| Hypersensitivity | Rash papulosquamous |
| Hypersensitivity | Rash pruritic |
| Hypersensitivity | Rash pustular |
| Hypersensitivity | Rash rubelliform |
| Hypersensitivity | Rash scarlatiniform |
| Hypersensitivity | Rash vesicular |
| Hypersensitivity | Reaction to azo-dyes |
| Hypersensitivity | Reaction to colouring |
| Hypersensitivity | Reaction to drug excipients |
| Hypersensitivity | Reaction to preservatives |
| Hypersensitivity | Red man syndrome |
| Hypersensitivity | Rhinitis allergic |
| Hypersensitivity | Scleral oedema |
| Hypersensitivity | Scleritis allergic |
| Hypersensitivity | Scrotal oedema |
| Hypersensitivity | Serum sickness |
| Hypersensitivity | Serum sickness-like reaction |
| Hypersensitivity | Shock |
| Hypersensitivity | Shock symptom |
| Hypersensitivity | Skin necrosis |
| Hypersensitivity | Skin reaction |
| Hypersensitivity | Skin test positive |
| Hypersensitivity | Solar urticaria |
| Hypersensitivity | Solvent sensitivity |
| Hypersensitivity | Stevens-Johnson syndrome |
| Hypersensitivity | Stoma site hypersensitivity |
| Hypersensitivity | Stoma site rash |
| Hypersensitivity | Swelling face |
| Hypersensitivity | Swollen tongue |
| Hypersensitivity | Tongue oedema |
| Hypersensitivity | Toxic epidermal necrolysis |
| Hypersensitivity | Toxic skin eruption |
| Hypersensitivity | Tracheal oedema |
| Hypersensitivity | Type I hypersensitivity |
| Hypersensitivity | Type II hypersensitivity |
| Hypersensitivity | Type III immune complex mediated reaction |
| Hypersensitivity | Type IV hypersensitivity reaction |
| Hypersensitivity | Urticaria |
| Hypersensitivity | Urticaria cholinergic |
| Hypersensitivity | Urticaria chronic |
| Hypersensitivity | Urticaria contact |
| Hypersensitivity | Urticaria papular |
| Hypersensitivity | Urticaria physical |
| Hypersensitivity | Urticaria pigmentosa |

Statistical Analysis Plan




| Category | PT |
|------------------|---------------------------|
| Hypersensitivity | Urticaria vesiculosa |
| Hypersensitivity | Vaginal exfoliation |
| Hypersensitivity | Vaginal ulceration |
| Hypersensitivity | Vasculitic rash |
| Hypersensitivity | Vessel puncture site rash |
| Hypersensitivity | Vulval ulceration |
| Hypersensitivity | Vulvovaginal rash |
| Hypersensitivity | Vulvovaginal ulceration |

Hyperphosphatemia: based on selected PTs below

| Category | PT |
|-------------------|----------------------------|
| Hyperphosphatemia | Hyperphosphatemia |
| Hyperphosphatemia | Blood phosphorus increased |
| Hyperphosphatemia | Blood phosphate abnormal |

Ectopic mineralization: based on a MedDRA search of 'calcification'

| Category | PT |
|-----------------------|---------------------------------|
| Ectopic calcification | Adrenal calcification |
| Ectopic calcification | Aortic calcification |
| Ectopic calcification | Aortic valve calcification |
| Ectopic calcification | Aortic valve sclerosis |
| Ectopic calcification | Articular calcification |
| Ectopic calcification | Bladder wall calcification |
| Ectopic calcification | Breast calcifications |
| Ectopic calcification | Bursa calcification |
| Ectopic calcification | Calcific deposits removal |
| Ectopic calcification | Calcification metastatic |
| Ectopic calcification | Calcification of muscle |
| Ectopic calcification | Calcinosis |
| Ectopic calcification | Calculus bladder |
| Ectopic calcification | Calculus prostatic |
| Ectopic calcification | Calculus ureteric |
| Ectopic calcification | Calculus urethral |
| Ectopic calcification | Calculus urinary |
| Ectopic calcification | Cardiac valve sclerosis |
| Ectopic calcification | Cerebral calcification |
| Ectopic calcification | Chondrocalcinosis |
| Ectopic calcification | Chondrocalcinosis pyrophosphate |
| Ectopic calcification | Cutaneous calcification |
| Ectopic calcification | Dystrophic calcification |
| Ectopic calcification | Heart valve calcification |




| Category | PT |
|-----------------------|-----------------------------------|
| Ectopic calcification | Heart valve stenosis |
| Ectopic calcification | Hepatic calcification |
| Ectopic calcification | Intervertebral disc calcification |
| Ectopic calcification | Intestinal calcification |
| Ectopic calcification | Ligament calcification |
| Ectopic calcification | Lymph node calcification |
| Ectopic calcification | Mitral valve calcification |
| Ectopic calcification | Mitral valve sclerosis |
| Ectopic calcification | Myocardial calcification |
| Ectopic calcification | Nephrocalcinosis |
| Ectopic calcification | Nephrolithiasis |
| Ectopic calcification | Ovarian calcification |
| Ectopic calcification | Pancreatic calcification |
| Ectopic calcification | Pericardial calcification |
| Ectopic calcification | Pleural calcification |
| Ectopic calcification | Prostatic calcification |
| Ectopic calcification | Pulmonary calcification |
| Ectopic calcification | Pulmonary valve calcification |
| Ectopic calcification | Pulmonary valve sclerosis |
| Ectopic calcification | Splenic calcification |
| Ectopic calcification | Stag horn calculus |
| Ectopic calcification | Tendon calcification |
| Ectopic calcification | Tracheal calcification |
| Ectopic calcification | Tricuspid valve calcification |
| Ectopic calcification | Tricuspid valve sclerosis |
| Ectopic calcification | Vascular calcification |

# Restless legs syndrome

| Category | PT |
|------------------------|---------------------------|
| Restless legs syndrome | Restless legs syndrome |
| Restless legs syndrome | Restlessness |
| Restless legs syndrome | Akathisia |
| Restless legs syndrome | Psychomotor hyperactivity |
| Restless legs syndrome | Sensory disturbance |
| Restless legs syndrome | Muscle cramp |
| Restless legs syndrome | Limb discomfort |
| Restless legs syndrome | Neuromuscular pain |
| Restless legs syndrome | Formication |